CLINICAL TRIAL: NCT05320094
Title: An Open-label Study to Evaluate the Effect of Activated Charcoal With Sorbitol on the Pharmacokinetics of Mavacamten in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Activated Charcoal With Sorbitol on the Single-dose of Mavacamten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV027-043
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: Mavacamten; Sorbitol; Activated Charcoal
MeSH Terms: conditions — Anthrax | interventions — MYK-461; Charcoal; Sorbitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mavacamten (Experimental)
  Interventions: Drug: Mavacamten
- Mavacamten and activated charcoal with sorbitol - Dose A (Experimental)
  Interventions: Drug: Mavacamten; Drug: Activated Charcoal with Sorbitol
- Mavacamten and activated charcoal with sorbitol - Dose B (Experimental)
  Interventions: Drug: Mavacamten; Drug: Activated Charcoal with Sorbitol

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
Drug: Activated Charcoal with Sorbitol — Specified dose on specified days
  Arms: Mavacamten and activated charcoal with sorbitol - Dose A; Mavacamten and activated charcoal with sorbitol - Dose B

SUMMARY:
The purpose of this study is to evaluate the effects of co-administration of activated charcoal with sorbitol on the single-dose drug levels of mavacamten in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kg/m^2, inclusive, at the Screening Visit
* Healthy, as determined by physical examination, vital signs, electrocardiograms (ECGs), and clinical laboratory assessments

Exclusion Criteria:

* Current or recent (within 3 months of study intervention administration) gastrointestinal disease
* History of sorbitol or fructose intolerance or inability to tolerate activated charcoal
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero extrapolated to infinite time ((AUC(INF)) | Up to 2 months
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration ((AUC(0-T)) | Up to 2 months
Maximum observed plasma concentration (Cmax) | Up to 1 month

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 3 months
Number of participants with serious adverse events (SAEs) | Up to 3 months
Number of participants with vital sign abnormalities exceeding predefined thresholds | Up to 3 months
Number of participants with electrocardiogram (ECG) abnormalities | Up to 3 Months
Number of participants with physical exam abnormalities | Up to 3 months
Number of participants with clinical laboratory evaluation abnormalities | Up to 3 months
Time of maximum observed plasma concentration (Tmax) | Up to 1 month
Apparent terminal plasma half-life (T-HALF) | Up to 2 months
Concentration at 24 hours (C24) | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Dallas, Texas, United States

REFERENCES:
- [Derived] Merali S, Chiang M, Sychterz C, Chao L, Simmons T, Xu Y, Zhao A, Attanasio M, Murthy B, Perera V. Effect of Activated Charcoal on Mavacamten Pharmacokinetics in Healthy Participants. Am J Cardiovasc Drugs. 2024 Jul;24(4):569-575. doi: 10.1007/s40256-024-00659-z. Epub 2024 Jun 26. PMID 38926266
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm